CLINICAL TRIAL: NCT05436613
Title: Community-based Transcranial Direct Current Stimulation Treatment for Bipolar Depression
Brief Title: Transcranial Direct Current Stimulation Therapy for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East London (Other)
Collaborators: University College, London (Other); King's College London (Other); Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Cynthia Fu, College Professor of Affective Neuroscience, University of East London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 308690
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Depression, Bipolar; Bipolar Disorder; Mood Disorders; Mental Disorder
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Mental Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device: transcranial direct current stimulation (Experimental): 6-week course of active tDCS treatment, consisting of 5 sessions per week for the first 3 weeks followed by 2 sessions per week for 3 weeks, for a total of 21 tDCS sessions. The duration of each session is 30 minutes.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — tDCS at 2mA in 30 minute sessions for 5 sessions per week for 3 weeks and then 2 sessions per week for 3 weeks.

SUMMARY:
Bipolar disorder is a severe and disabling disorder. The course of illness is often progressive but is highly heterogeneous between individuals and within the lifetime for an individual. The most common treatments are medications. However, for many individuals, combinations of medications are often required, and full recovery is infrequent.

The novel brain stimulation treatment, transcranial direct current stimulation (tDCS), is a potential first-line treatment for bipolar depression. The present research question is whether tDCS can be provided as a home-based treatment for bipolar depression for adults with bipolar disorder.

DETAILED DESCRIPTION:
The novel brain stimulation treatment, transcranial direct current stimulation (tDCS), is a potential first-line treatment for bipolar disorder. tDCS generates a small electric current which modulates how easy it is for active brain cells to discharge. The device is a headband worn over the forehead with two electrodes, which are small metal discs, where the current comes from. tDCS does not directly stimulate brain cells to cause a seizure like electroconvulsive therapy (ECT) and it does not induce brain cells to discharge like transcranial magnetic stimulation (TMS).

Clinical studies have shown that tDCS treatment could help to improve the symptoms of depression. The main side effects have been redness, skin irritation or sensations (itching, tingling or burning) under the electrodes. Less commonly reported side effects include headache or tiredness. tDCS is a portable and safe treatment.

The studies to date have mostly looked at tDCS treatment which has been provided in a research setting. This is a problem because the treatment requires daily sessions for several weeks which could limit whether individuals would be able to go every day. As tDCS is a portable and safe treatment, it could be provided in the community.

The present study is a proof-of-concept trial to assess the efficacy, acceptability and safety of tDCS treatment for bipolar depression within a community-based setting.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar disorder based on DSM-5 criteria
* minimum score of 18 on the MADRS
* being on a stable dosage of mood stabilizing medication for a minimum of two weeks

Exclusion Criteria:

* comorbid psychiatric disorder
* significant risk of suicide or self harm
* any contraindications to tDCS, including implanted electronic medical devices
* history of epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Fu, MD, PhD, Principal Investigator — University of East London
Locations (1):
- University of East London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mutz J, Edgcumbe DR, Brunoni AR, Fu CHY. Efficacy and acceptability of non-invasive brain stimulation for the treatment of adult unipolar and bipolar depression: A systematic review and meta-analysis of randomised sham-controlled trials. Neurosci Biobehav Rev. 2018 Sep;92:291-303. doi: 10.1016/j.neubiorev.2018.05.015. Epub 2018 May 12. PMID 29763711
- [Background] Mutz J, Vipulananthan V, Carter B, Hurlemann R, Fu CHY, Young AH. Comparative efficacy and acceptability of non-surgical brain stimulation for the acute treatment of major depressive episodes in adults: systematic review and network meta-analysis. BMJ. 2019 Mar 27;364:l1079. doi: 10.1136/bmj.l1079. PMID 30917990
- [Background] Woodham R, Rimmer RM, Mutz J, Fu CHY. Is tDCS a potential first line treatment for major depression? Int Rev Psychiatry. 2021 May;33(3):250-265. doi: 10.1080/09540261.2021.1879030. Epub 2021 Mar 11. PMID 33706656
- [Background] Woodham RD, Rimmer RM, Young AH, Fu CHY. Adjunctive home-based transcranial direct current stimulation treatment for major depression with real-time remote supervision: An open-label, single-arm feasibility study with long term outcomes. J Psychiatr Res. 2022 Sep;153:197-205. doi: 10.1016/j.jpsychires.2022.07.026. Epub 2022 Jul 8. PMID 35839661
- [Derived] Rezaei H, Woodham RD, Ghazi-Noori AR, Ritter P, Bauer M, Young AH, Bramon E, Fu CHY. Acceptability of home-based transcranial direct current stimulation (tDCS) in bipolar depression: thematic analysis of individual views. BMC Psychiatry. 2025 May 26;25(1):549. doi: 10.1186/s12888-025-06948-4. PMID 40420071
- [Derived] Rezaei H, Woodham RD, Ghazi-Noori AR, Ritter P, Bauer M, Young AH, Bramon E, Fu CHY. Acceptability of Home-Based Transcranial Direct Current Stimulation (tDCS) in Bipolar Depression: Thematic Analysis of Individual Views. Res Sq [Preprint]. 2025 Apr 15:rs.3.rs-5967699. doi: 10.21203/rs.3.rs-5967699/v1. PMID 40321750
- [Derived] Ghazi-Noori AR, Woodham RD, Rezaei H, Sharif MS, Bramon E, Ritter P, Bauer M, Young AH, Fu CHY. Home-based transcranial direct current stimulation in bipolar depression: an open-label treatment study of clinical outcomes, acceptability and adverse events. Int J Bipolar Disord. 2024 Aug 20;12(1):30. doi: 10.1186/s40345-024-00352-9. PMID 39162912

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device: Transcranial Direct Current Stimulation
Started | 44
Completed | 32
Not Completed | 12
Not completed — Lost to Follow-up | 9
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Device: Transcranial Direct Current Stimulation
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.27 (12.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 44
Ammons Quick Test (measure of IQ) [Mean (Standard Deviation); unit: units on a scale] — The Ammons Quick Test is a measure of receptive vocabulary, verbal intelligence, and verbal information processing.
  Range of scores representing Intelligence Quotient (IQ) - 40 to 135. Higher values indicate higher IQ, or greater intelligence.
  units on a scale | 100.66 (9.29)
MADRS: Montgomery-Åsberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — MADRS is a clinician rated diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  Range of scores: 0 to 60. Higher scores represent greater severity of depressive symptoms.
  units on a scale | 24.59 (2.64)
HDRS-17: Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — HDRS-17 is a clinician rated diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  Range of scores: 0 to 52. Higher scores represent greater severity of depressive symptoms.
  units on a scale | 19.98 (2.62)
HAMA: Hamilton Anxiety Rating Scale [Mean (Standard Deviation); unit: units on a scale] — HAMA is a clinician rated diagnostic questionnaire used to measure the severity of anxiety symptoms in patients with mood disorders.
  Range of scores: 0 to 56. Higher scores represent greater severity of anxiety symptoms.
  units on a scale | 16.55 (5.26)
YMRS: Young Mania Rating Scale [Mean (Standard Deviation); unit: units on a scale] — YMRS is a clinician rated diagnostic questionnaire used to measure the severity of manic symptoms in patients with mood disorders.
  Range of scores: 0 to 60. Higher scores represent greater severity of manic symptoms.
  units on a scale | 2.20 (1.49)
PHQ-9: Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — PHQ-9 is a self-reported diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders.
  Range of scores: 0 to 27. Higher scores represent greater severity of depressive symptoms.
  units on a scale | 16.80 (4.94)
SDS: Sheehan Disability Scale [Mean (Standard Deviation); unit: units on a scale] — SDS is a brief, self -report questionnaire designed to assess functional impairment caused by psychiatric or medical symptoms across three key life domains: work/school, social life/leisure activities, and family life/home responsibilities.
  Scores range from 0 to 30 with higher scores indicating greater functional impairment.
  units on a scale | 20.77 (5.87)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response [ Time Frame: At 6 Weeks Following Course of tDCS Treatment ]
Description: As measured by clinician-rated Montgomery Asberg Depression Rating Scale (MADRS) score improvement of 50% or more from baseline following the course of tDCS treatment.
Time Frame: 6 weeks
Population: Intention to Treat analysis including all participants who enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Transcranial Direct Current Stimulation
Number analyzed (Participants) | 44
Participants | 34

2. Secondary Outcome: Participant Retention at the End of the Treatment
Description: The number of participants who have completed a minimum of 15 tDCS sessions
Time Frame: 6 weeks (visit 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Transcranial Direct Current Stimulation
Number analyzed (Participants) | 44
Participants | 41

3. Secondary Outcome: Participant Acceptability Questionnaire Scales
Description: Participants were asked how acceptable they found the tDCS treatment after the 6-week course of treatment. They were given responses on a 7-point Likert style scale. The number of participants who rated the tDCS treatment as acceptable on the Treatment Acceptability Questionnaire (Likert responses 5, 6 or 7) are reported.
Time Frame: Week 6 (Visit 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Transcranial Direct Current Stimulation
Number analyzed (Participants) | 41
Participants | 41

4. Other Pre Specified Outcome: MADRS Remission Rate
Description: Trained rater measure of depressive symptoms: Montgomery-Åsberg Depression Rating Scale (MADRS) remission rate: a score of less than 10 following the course of tDCS
Time Frame: 6 weeks (Visit 21)
Measure: Count of Participants; unit: Participants
Arm/Group | Device: Transcranial Direct Current Stimulation
Number analyzed (Participants) | 44
Participants | 21

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Adverse events reported during the trial
Arm/Group | Device: Transcranial Direct Current Stimulation
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Transcranial Direct Current Stimulation (N=44)
Throat Infection (Immune system disorders) | 1 (1) — Requiring hospitalisation not related to the study intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Transcranial Direct Current Stimulation (N=44)
Headache (Nervous system disorders) | 9 (22)
Scalp pain (Skin and subcutaneous tissue disorders) | 5 (24)
Tingling (Skin and subcutaneous tissue disorders) | 43 (716)
Itching (Skin and subcutaneous tissue disorders) | 10 (252)
Burning sensation (Skin and subcutaneous tissue disorders) | 34 (226)
Skin redness (Skin and subcutaneous tissue disorders) | 34 (347)
Trouble concentrating (Nervous system disorders) | 2 (6)
Sleepiness (Nervous system disorders) | 9 (25)
Acute mood change (Nervous system disorders) | 4 (7)
Sore feeling at electrode site (Skin and subcutaneous tissue disorders) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT05436613/Prot_SAP_000.pdf